CLINICAL TRIAL: NCT06535243
Title: Evaluation of the Efficacy of "Lifespan Integration" Therapy in Patients With Complex Post-Traumatic Stress Disorder
Brief Title: Evaluation of the Efficacy of "Lifespan Integration" (LI) Therapy in Patients With Complex Post-Traumatic Stress Disorder
Acronym: EVALI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Principal Investigator, Alexandru GAMAN, Medic Doctor MD, Centre Hospitalier St Anne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D21-P019
Record Dates: First submitted 2024-04-28; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Post-Traumatic Stress Disorder Complex; Psychiatric Disorder; Abuse Neglect; Abuse Physical; Abuse, Sexual; Abuse Domestic; Abuse Verbal
Keywords: Lifespan Integration Therapy; Psychotrauma type II; Abuse; Victims; Complex Post-traumatic Stress Disorder; Psychotherapy
MeSH Terms: conditions — Mental Disorders; Coitus

STUDY DESIGN:
Intervention Model Description: eligible candidates to be included in this cohort should be
  * older than 18 yo
  * French speaking
  * with a diagnosis of complex PTSD as confirmed by 1/clinical interview with a trained psychiatrist and 2/ scores for the International Trauma Questionnaire (ITQ), clinical tool based on the ICM 11 criteria
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LI Therapy (Experimental): LI Therapy will be delivered in two recruiting centers by experienced LI Therapy trained psychologists or psychiatrists (a minimum level three of training is required) The intervention will consist in delivering 15 "Basic" Protocol therapy sessions targeting symptoms of complex PTSD The study contains one single arm. One extra-session called PTSD protocol could be optionally delivered if the patient had a very recent trauma that could exacerbate his PTSD symptoms. This session is delivered in the beginning of the research protocol.
  Interventions: Behavioral: Lifespan Integration Therapy (LI)

INTERVENTIONS:
Behavioral: Lifespan Integration Therapy (LI) — same as above

SUMMARY:
The study aims to evaluate the efficacy of a relatively new type of psychotherapy called Lifespan Integration (LI) in patients suffering of complex PTSD

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with complex PTSD
* French speaking
* first time following an LI type of therapy
* psychotropic treatment is allowed

Exclusion Criteria:

* no other parallel psychotherapy is accepted (if the patient underwent recently any other type of psychotherapy, a "wash out " period of minimum 4 weeks is required )
* no active manic episode at the time of inclusion
* no active psychotic episode at the time of inclusion
* no chronic psychotic disorder diagnosis
* no autistic spectrum disorder diagnosis ,
* no intellectual deficit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
change of the scores of International Trauma Questionnaire | maximum one year
  International Trauma Questionnaire measures subscores of simple and complex PTSD, the score is calculated using an algorithm, a minimum score of 8 for the PTSD simple part and of 8 for PTSD complex part is needed in order to diagnose a complex PTSD; the maximum score for simple PTSD is 16, same for complex PTSD.

SECONDARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) Score | maximum one year
  the DERS scale (Gratz and Roemer, 2004) contains 36 Likert Scale questions with scores from 1 to 5; the scale can generate a total score and six underscores (assessing nonacceptance, goals, impulse, awareness, strategies, clarity); in a general population cohort the mean score was of 77.99 (SD= 20.72) for N=260 women and 80.66 (SD= 18.79) for N=97 men

OTHER OUTCOMES:
Rosenberg Self - Esteem Scale (RSES) (Rosenberg, 1965) | maximum one year
  RSES is one of the most widely used measures of global self esteem; it contains 10 questions with answers ranging from 0 (poor) to 3 (excellent); five questions are positively worded and five questions are negatively worded. Sinclair and colleagues, 2010 reported a mean score of 22.62 (SD=5.80) in a general population cohort from the US of N=503 individuals

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru GAMAN, MD, Principal Investigator — GHU Paris Hôpital St Anne
Locations (1):
- CHU St Anne, Paris, Île-de-France Region, France